CLINICAL TRIAL: NCT05713734
Title: Bleeding of Unknown Cause, Insight Into a Multifactorial Bleeding Disorder: a Swiss Case-control Study
Brief Title: Bleeding of Unknown Cause: a Swiss Case-control Study
Acronym: SWISS-BUC
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Casini Alessandro, Principal investigator, University Hospital, Geneva
Other Study IDs: CCER 2022-02121
Record Dates: First submitted 2023-01-27; First posted 2023-02-06 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Bleeding Disorder
Keywords: Bleeding; Hemostatics; Fibrin; Fibrinolysis; Thrombin
MeSH Terms: conditions — Hemostatic Disorders; Hemorrhage | interventions — Fibrinolysis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma and EDTA samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Patients with bleeding of unknown cause
  Interventions: Diagnostic Test: Thrombin generation; Diagnostic Test: Fibrinolysis; Diagnostic Test: Fibrin clot structure; Diagnostic Test: Coated platelets
- Controls: Healthy voluntaries without bleeding tendency
  Interventions: Diagnostic Test: Thrombin generation; Diagnostic Test: Fibrinolysis; Diagnostic Test: Fibrin clot structure; Diagnostic Test: Coated platelets

INTERVENTIONS:
Diagnostic Test: Thrombin generation — Measurement of thrombin generation by ST Genesia
Diagnostic Test: Fibrinolysis — Measurement of fibrinolysis by Lysis Timer
Diagnostic Test: Fibrin clot structure — Measurement of fibrin polymerisation and permeability
Diagnostic Test: Coated platelets — Measurement of coated platelets by flow cytometry

SUMMARY:
The goal of this prospective cohort is to identified specific biological patterns in patients with a bleeding of unknown cause and to study the specific mechanisms of the bleeding disorder for each subset of patients.

DETAILED DESCRIPTION:
Patients with bleeding of unknown cause are included. At baseline, blood will be drawn to evaluate the hemostatic profile. Findings are compared to a control group of healthy individuals. Patients and controls are followed for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Man with ISTH BAT>3. If the calculated score includes a surgical bleeding, then two other items of the score should be >0
* Woman with ISTH BAT >5 points. If the calculated score includes a surgical or a postpartum bleeding, then two other items of the score should be >0

Exclusion Criteria:

* Ongoing pregnancy
* Intake of antithrombotic treatment or non-steroidal anti-inflammatory drugs for least 10 days at time of blood collection
* Intake of antifibrinolytic or blood product administration (factor concentrate, frozen fresh plasma, prothrombin complex concentrate) for least 14 days before blood collection
* Active cancer (defined as cancer diagnosis within the last five years or treatment within the two last years before study inclusion)
* Active autoimmune disease
* Active chronic inflammatory disease
* Severe liver disease (cirrhosis > Child A)
* Renal insufficiency stage 3
* Active or recent infection (within the last 30 days)
* Recent hospitalization (<3 months)
* Recent surgery (<3 months)
* Recent trauma requiring medical intervention (<3 months)

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Women and men aged 16-65 years who have been diagnosed as patients with bleeding of unknown cause Women and men aged 16-65 years without bleeding tendency
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Fibrin clot polymerisation | At inclusion
  maximal absorption (optical density)
Fibrin clot permeability | At inclusion
  darcy coefficient (ks, cm2)
Fibrinolysis | At inclusion
  Clot lysis time (min)
Thrombin generation | At inclusion
  Endogenous thrombin potential (ETP, nM x min)
Coated platelets | At inclusion
  Absolute number of coated platelets

SECONDARY OUTCOMES:
Fibrinogen gamma' levels | At inclusion
  Ratio fibrinogen gamma'/total fibrinogen (%)
Scan electron microscopy | At inclusion
  Fibrin fiber diameter (nm)
Clot retraction | At inclusion
  Ratio clot weight/serum extruded (%)
Plasmin generation | At inclusion
  Plasmin (nM)
Fibrin clot formation (thrombodynamics) | At inclusion
  Initial rate of clot growth (μM/min)
Major bleeding episodes | Three years
  Incidence of major bleeding
Non-major bleeding episodes | Three years
  Incidence of clinically relevant non-major bleeding
Health related quality of life | three years
  SF36 questionnaire, 0 - 100 (high score, better outcome)
International Society Thrombosis Hemostasis Bleeding assessment tool | three years
  ISTH BAT score, 0 - 56 (high score, worse outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Casini, Principal Investigator — University Hospitals of Geneva
Locations (7):
- Switzerland (7):
  - Ospedale Regionale di Bellinzona, Bellinzona
  - Inselspital - Universitätsspital Bern, Bern
  - University Hospital, Geneva
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Gruppo Ospedaliero Moncucco, Lugano
  - Kantonsspital St.Gallen, Sankt Gallen
  - USZ - Universitätsspital Zürich, Zurich